CLINICAL TRIAL: NCT06250764
Title: Investigation the Relationship Between Periodontal Disease and 'Asprosin, Adropin, Irisin' Levels
Brief Title: Asprosin, Adropin, Irisin Levels in Periodontitis
Status: Completed | Type: Observational
Sponsor: AYSAN LEKTEMUR ALPAN (Other)
Responsible Party: Sponsor-Investigator, AYSAN LEKTEMUR ALPAN, Associate Professor, Pamukkale University
Organization: Pamukkale University (Other)
Other Study IDs: 2020/9-10
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Periodontal Diseases; Gingivitis; Obesity
Keywords: adropin; asprosin; irisin; periodontal disease; gingival crevicular fluid
MeSH Terms: conditions — Periodontal Diseases; Gingivitis; Obesity; Arachnodactyly

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- GROUP 1 (periodontally healthy ): An individual to be considered to have periodontal health according to this definition, the percentage of sites with bleeding on probing should be no more than 10%, and the probing depth should be 3 mm or less
  Interventions: Diagnostic Test: Clinical periodontal measuremenets; Diagnostic Test: ELISA test from gingival crevicular fluid (GCF)
- GROUP 2 (gingivitis): Patients with gingivitis had PD ≤3 mm, BOP in ≥30% of the probing sites, and no interproximal AL or radiographic bone loss
  Interventions: Diagnostic Test: Clinical periodontal measuremenets; Diagnostic Test: ELISA test from gingival crevicular fluid (GCF)
- GROUP 3(generalized stage I and stage II periodontitis): Stage I periodontitis was diagnosed with interdental attachment loss (AL) ranging between 1 and 2 mm at the site of greatest loss. Radiographic bone loss (BL) is limited to less than 15% and no tooth loss. Additionally, the maximum probing depth (PD) is equal to or less than 4 mm or primarily involves horizontal bone loss. Stage II periodontitis was diagnosed with interdental attachment loss (AL) is ranging between 3 and 4 mm at the site of greatest loss. Radiographic bone loss (BL) extends to a range of 15% to 33%, there is no tooth loss. The maximum probing depth (PD) is equal to or less than 5 mm or primarily involves horizontal bone loss.
  Interventions: Diagnostic Test: Clinical periodontal measuremenets; Diagnostic Test: ELISA test from gingival crevicular fluid (GCF)
- GROUP 4 (generalized stage III and stage IV periodontitis): Stage III periodontitis is diagnosed with interdental attachment loss (AL) is ≥ 5, radiographic bone loss (BL) extends to mid-third of the root and beyond, tooth loss may become evident ≤4 teeth. Either PD ≥ 6 mm or vertical BL ≥ 3 mm, or Class II/III furcation involvement, or moderate ridge defect. Stage IV periodontitis is diagnosed with interdental attachment loss (AL) is ≥ 5 mm at the site of greatest loss, radiographic BL extending to mid-third of the root and beyond. ≥5 tooth loss due to periodontitis is evident. In addition to Stage III, either masticatory dysfunction, or secondary occlusal trauma (tooth mobility degree ≥ 2), or severe ridge defect, or bite collapse, or teeth drifting and flaring
  Interventions: Diagnostic Test: Clinical periodontal measuremenets; Diagnostic Test: ELISA test from gingival crevicular fluid (GCF)

INTERVENTIONS:
Diagnostic Test: Clinical periodontal measuremenets — The periodontal assessment was performed by a single trained examiner (S.D.). A graded periodontal probe (Williams, Hu-Friedy, Chicago, IL, USA) was used to measure probing depth (PD) which was determined as the depth from the gingival margin to the bottom of the gingival sulcus/periodontal pocket, clinical attachment loss (CAL) which was calculated as the distance from the cemento-enamel junction to the bottom of the periodontal pocket and dual recording (+/-) of bleeding on probing (BOP), gingival index (GI) and plaque index (PI) in total except third molars G
Diagnostic Test: ELISA test from gingival crevicular fluid (GCF) — GCF sampled from the buccal aspects of non-contiguous proximal regions in maxillary single-rooted teeth. In the periodontitis groups, fluid samples were taken from the two deepest pockets. In the gingivitis and periodontal healthy groups, fluid samples were obtained from areas with and without visible inflammation, respectively

SUMMARY:
The recently discovered association of the hormones 'asprosin, adropin and irisin' with obesity and metabolic status, as well as the fact that periodontal diseases are affected by obesity and nutrition bilaterally, have led us to investigate the relationship between selected target markers and periodontal disease. The primary aim and main objective of this study is to increase the knowledge and to direct future researches as a result of the lack of adequate research in the past and the very limited investigations with these hormones in dentistry and periodontology.

Our study was conducted on 122 patients who applied to Adıyaman University Faculty of Dentistry and were referred to the Department of Periodontology for routine periodontal controls. Participants' gender, age, height, weight, BMI, education level, tooth brushing and flossing habits as well as clinical parameters PI, GI, SCD, CAS and SDI were noted. Participants were divided into 4 groups as healthy, gingivitis, initial periodontitis and advanced periodontitis and grouped according to the current periodontal classification of 2017. DOS was collected from the groups for examination and 'asprosin, adropin and irisin' values in the samples were evaluated by ELISA test.

DETAILED DESCRIPTION:
A total of 122 patients participated in the study. All patients participating in the trial received written and verbal information about the purpose and method of the study and signed consent. Patients with cardiovascular disease, liver and kidney disease, metabolic disorders, diabetes, asthma, thyroid dysfunction, who used antibiotics or anti-inflammatory drugs within the last three months, who received periodontal treatment within the last six months, obese patients with body mass index (BMI) ≥ 30 kg/m2 according to the reference range determined by the World Health Organization, and patients who refused to participate were excluded from the study. In order to calculate the BMI of the individuals included in the study, height-weight information, tooth brushing frequency in order to determine oral hygiene habits, and educational status were also recorded to determine economic levels. Age and gender were also noted. Individuals aged 25-60 years were divided into four groups according to their periodontal status.

The periodontal assessment was performed by a single trained examiner (S.D.). A graded periodontal probe (Williams, Hu-Friedy, Chicago, IL, USA) was used to measure probing depth (PD), which was determined as the depth from the gingival margin to the bottom of the gingival sulcus/periodontal pocket; clinical attachment loss (CAL) which was calculated as the distance from the cemento-enamel junction to the bottom of the periodontal pocket and dual recording (+/-) of bleeding on probing (BOP), gingival index (GI) and plaque index (PI) in total except third molars. To assess the intra-examiner calibration, Cronbach's alpha was used and its value was 0.90 for PD and CAL measures. Alveolar bone loss (ABL) was determined in each participant by orthopantomography. The distance between the cemento-enamel junction and the bone crest was measured in both mesial and distal regions and its ratio to the root length was calculated to assess bone loss. The periodontal status of the patients was evaluated based on the Classification of Periodontal and Peri-Implant Diseases and Conditions from the 2017 World Workshop. Participants were classified into four distinct groups based on their periodontal conditions:

1. Group 1: 30 periodontally healthy individuals;
2. Group 2: 30 patients with gingivitis;
3. Group 3: 32 patients with generalized stage I and stage II periodontitis;
4. Group 4: 30 patients with generalized stage III and stage IV periodontitis. An individual to be considered to have periodontal health according to this definition, the percentage of sites with bleeding on probing should be no more than 10%, and the probing depth should be 3 mm or less. Patients with gingivitis had PD ≤3 mm, BOP in ≥30% of the probing sites, and no interproximal AL or radiographic bone loss. Stage I periodontitis was diagnosed with interdental attachment loss (AL) ranging between 1 and 2 mm at the site of greatest loss. Radiographic bone loss (BL) is limited to less than 15% and no tooth loss. Additionally, the maximum probing depth (PD) is equal to or less than 4 mm, which primarily involves horizontal bone loss. Stage II periodontitis was diagnosed with interdental attachment loss (AL) ranging between 3 and 4 mm at the site of greatest loss. Radiographic bone loss (BL) extends to a range of 15% to 33%; there is no tooth loss. The maximum probing depth (PD) is equal to or less than 5 mm, or primarily involves horizontal bone loss. Stage III periodontitis is diagnosed when interdental attachment loss (AL) is ≥ 5, radiographic bone loss (BL) extends to the mid-third of the root and beyond, and tooth loss may become evident ≤4 teeth. Either PD ≥ 6 mm or vertical BL ≥ 3 mm, or Class II/III furcation involvement, or moderate ridge defect. Stage IV periodontitis is diagnosed with interdental attachment loss (AL) of ≥ 5 mm at the site of greatest loss, with radiographic BL extending to the mid-third of the root and beyond. ≥5 tooth losses due to periodontitis are evident. In addition to Stage III, either masticatory dysfunction, secondary occlusal trauma (tooth mobility degree ≥ 2), severe ridge defect, bite collapse, or teeth drifting and flaring

ELIGIBILITY:
Inclusion Criteria:

All patients but exclusion criteria

Exclusion Criteria:

Patients with cardiovascular disease, liver and kidney disease, metabolic disorders, diabetes, asthma, thyroid dysfunction, who used antibiotics or anti-inflammatory drugs within the last three months, who received periodontal treatment within the last six months, obese patients with body mass index (BMI) ≥ 30 kg/m2 according to the reference range determined by the World Health Organisation, and patients who refused to participate were excluded from the study

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients admitted to the periodontology clinic between the study dates
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Association of PD and adipokine values | only baseline measurement the patients were seen once
  correlation identification using SPSS between pocket depth and these adipokines in periodontitis patients

CONTACTS AND LOCATIONS:
Overall Officials: METİN ÇALIŞIR, PHD, Principal Investigator — Adiyaman University; Sevde DEMİRCİ, Study Director — Adiyaman University
Locations (1):
- Adıyaman University Faculty of Dentistry, Adıyaman, Turkey (Türkiye)

REFERENCES:
- [Background] Loesche WJ, Grossman NS. Periodontal disease as a specific, albeit chronic, infection: diagnosis and treatment. Clin Microbiol Rev. 2001 Oct;14(4):727-52, table of contents. doi: 10.1128/CMR.14.4.727-752.2001. PMID 11585783
- [Background] Torumtay Cin G, Fenkci SM, Kilic ID, Aslan HS, Sevgican CI, Senol H. The effects of severe periodontitis on arterial stiffness using cardio-ankle vascular index in patients with type 2 diabetes. J Periodontal Res. 2024 Feb;59(1):74-83. doi: 10.1111/jre.13202. Epub 2023 Nov 1. PMID 37909328